CLINICAL TRIAL: NCT02239458
Title: DPP-IV Inhibition Prior to Development of Diabetes in Patients With Cystic Fibrosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ram Weiss (Other)
Responsible Party: Sponsor-Investigator, Ram Weiss, Head of the Department of Human Metabolism and Nutrition, Hadassah Medical Organization
Organization: Hadassah Medical Organization (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 0388-14-HMO
Record Dates: First submitted 2014-09-08; First posted 2014-09-12 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2014-09

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — saxagliptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Placebo (Placebo Comparator): Placebo intake during 3 months
- Saxagliptin 5mg (Active Comparator): Saxagliptin dose of 5mg for 3 months
  Interventions: Drug: Saxagliptin

INTERVENTIONS:
Drug: Saxagliptin
  Other Names: Onglyza
  Arms: Saxagliptin 5mg

SUMMARY:
Cystic fibrosis related diabetes (CFRD) is a common co-morbidity in patients with CF. The underlying pathophysiology of cystic fibrosis related diabetes (CFRD) is still a matter of investigation. In addition to localized tissue damage developing similar to that of the exocrine pancreas, other mechanisms may be involved. We have shown that a potential contributing factor to the patho-physiology of CFRD may be an abnormal gut derived hormonal profile, specifically of lower incretin hormone responses, prior to development of CFRD.

We propose that an altered incretin response, probably due to impaired interaction of nutrients with the gut mucosa due to thickened secretions, may play a role in the development of the disease. Specifically, low GIP and GLP-1, may explain the poor β-cell function observed in these patients prior to CFRD appearance. These incretins have known trophic effects on β-cells, and thus their lower levels may contribute to the development of quantitative as well as qualitative defects in β-cell function and thus may lead to the development of CFRD. Thus, increasing levels of these incretins using a DPP-IV inhibitor may improve glucose metabolism and delay/prevent the development of CFRD.

We hypothesize that Saxagliptin will increase the oDI compared to placebo and will thus provide relative protection from diabetes development and in addition we expect that Saxagliptin will lead to overall increased insulin concentrations and thus shift the metabolic milieu to a more anabolic state. This will manifest as weight gain and reduction in inflammation.

DETAILED DESCRIPTION:
The following proposal includes testing the utility of DPP-IV inhibition in adult patients with CF without CFRD. This will be achieved by a randomized double blind controlled trial of Saxagliptin 5 mg vs. placebo which will be performed for 3 months in 60 patients with CF without CFRD. The study will be for 3 months of use and will consist of two arms:

1. Saxagliptin 5mg
2. Placebo. the primary outcome of this study will be the oral disposition index oDI , derived from the OGTT. The oDI has been shown across age groups and metabolic phenotypes to be an excellent predictor of diabetes development over time . We postulate that Saxagliptin will increase incretin concentrations and thus improve insulin secretion. This will manifest as an increased oral disposition index (oDI), reflecting an improved beta cell response in the context of prevailing insulin sensitivity. The oDI is a useful predictor of diabetes development over time and its increase will provide evidence for protection from diabetes in this special study population

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* Diagnosis of CF
* No CFRD on baseline OGTT
* Normal kidney function
* No history of pancreatitis
* Able and willing to consent and participate

Exclusion Criteria:

* Acute illness/exacerbation of CF associated lung disease
* Receiving immune-modulators following lung/pancreas transplant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Oral Disposition Index | The ODI will be calculated at baseline (Day 1) and at End point (day 90- 3 months)
  The oDI is a useful predictor of diabetes development over time and its increase will provide evidence for protection from diabetes in this special study population

CONTACTS AND LOCATIONS:
Overall Officials: Eitan Kerem, MD, Principal Investigator — Hadassah Ein Kerem
Locations (1):
- Hadassah Ein Kerem/Har Hazofim, Jerusalem, Israel